CLINICAL TRIAL: NCT07129369
Title: Evaluating the Effects of a Peer-facilitated, Acceptance-based Self-learning for Illness Management (PASIM) Program for Adults With Recent-onset Psychosis: A Randomized Controlled Trial
Brief Title: Effects of a Peer-facilitated, Acceptance-based Self-learning for Illness Management (PASIM) Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Integrated Community Centers for Mental Wellness (Unknown); Psychiatric outpatient clinics (Unknown)
Responsible Party: Principal Investigator, Prof. Wai Tong CHIEN, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 14608525
Record Dates: First submitted 2025-08-06; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Psychotic Disorders; Recent-Onset Psychosis
Keywords: Randomized controlled trial; Acceptance-based intervention; Peer support; Self help; Recent-onset psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Center / Clinical staff
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PASIM group (Experimental): Participants in the PASIM program will study and complete the self-learning manual (printed and online versions available) with 5 modules for ROP patients (translated, refined and validated by research team) and participate in 4 group sessions facilitated by a peer-support worker over 5 months.
  Interventions: Behavioral: PASIM program; Behavioral: Usual-Care-only
- Psychoeducation group (Experimental): The psychoeducation group (12 two-hour sessions, 5 subgroups with 12-14 patients per group) will be led by one trained psychiatric nurse experienced in psychiatric rehabilitation and psychoeducation group.
  Interventions: Behavioral: Psychoeducation; Behavioral: Usual-Care-only
- Usual-care-only group (Other): This control group (and 2 intervention groups) will receive usual community mental healthcare services provided by POPCs and ICCMWs. Patients in ICCMWs and POPCs may receive services in commons, including occupational/living skills training, education on psychosis care, recreational services, and individual and/or family counseling and referrals to social and health care services as needed. The control group will also receive an information booklet about illness self-care to minimize the Hawthorne effect from the PASIM manual reading.
  Interventions: Behavioral: Usual-Care-only

INTERVENTIONS:
Behavioral: PASIM program — The program consists of 5 modules for ROP patients (translated, refined and validated by research team) and 4 group sessions (1.5 hours per session; 8-10 members/group; in-between completion of the 5 modules) facilitated by a peer-support worker over 5 months. The 5 modules include: Module 1-Patient's well-being; Module 2-Getting the best out of support services; Module 3-Acceptance and insight toward psychosis and long-term self-care; Module 4-Dealing with psychosocial effects of the illness- I; and Module 5-Dealing with physical/mental health effects of the illness- II. The 4 group sessions will be conducted at the orientation and after reading the 1st, 3rd and 5th module to introduce the program, encourage to complete the module per month, performing value clarifying and acceptance (psychological flexibility) exercises, and clarify and discuss self-care learning and and challenges.
  Arms: PASIM group
Behavioral: Psychoeducation — The psychoeducation group (5 subgroups with 12-14 patients per group) will be led by one trained psychiatric nurse experienced in psychiatric rehabilitation and psychoeducation group. The program consists of 12 two-hour sessions held weekly or biweekly (similar to the PASIM) over 5 months with four key components, including introduction and goal setting; an education workshop on psychosis care and community service; learning effective coping and self-care skills with rehearsals/reviews; and skills practices and preparing for future life.
  Arms: Psychoeducation group
Behavioral: Usual-Care-only — Participants receive usual community mental healthcare services provided by POPCs and ICCMWs.

SUMMARY:
Psychosis is a very disabling mental illness with a wide range of dysregulations and disruptions in cognition, emotions, and behaviors, resulting in poor functioning and frequent relapses, especially in the first five years of the illness. There is a knowledge gap about whether Peer-facilitated, Acceptance-based Self-learning for Illness Management (PASIM) can have longer-term and more significant benefits than current professional-led psychoeducation in diverse health outcomes of these psychotic patients such as functioning, problem-solving, and recovery. This multi-center randomized controlled trial with repeated measures, 3-arm design is proposed to test and compare the effects between two alternative interventions (PASIM and Psychoeducation Group program) and a usual-care-only group over an 18-month follow-up.

DETAILED DESCRIPTION:
Objectives:

To test the primary hypothesis that the PASIM program can produce significantly greater improvements than psychoeducation and/or usual-care only groups at 1-week, 9-month, and/or 18-month follow-ups on patients' functioning; To test the hypothesis that the PASIM program will produce significantly greater improvements than psychoeducation and usual-care-only over the 18-month follow-ups in patients' psychotic symptoms, problem-solving, illness insight, rehospitalization rates, and/or service satisfaction (secondary outcomes); To explore the strengths, weaknesses and areas for improvements of and satisfaction with the PASIM program, from participants' and peer facilitators' perspectives, using individual semi-structured interviews.

Design: A multi-center randomized controlled trial with repeated measures, 3-arm design will be conducted with both outcome and process evaluation.

Subjects: 186 adults with recent-onset psychosis and randomly assigned into three study groups.

Data collection procedure: After explaining the study and ethical issues to participants, written consent and then baseline measurement will be obtained. During interventions, participants' attendance, workbook completion and attritions will be monitored. At 1-week (Posttest-1), and 9- (Posttest-2) and 18-month (Posttest-3) post-intervention, outcome measurements will be evaluated. In addition, individual semi-structured interviews will be conducted after Posttest-1.

Data analysis: Generalized Estimating Equation test will be used to compare mean-value changes in individual outcomes, and Kaplan-Meier survival-analysis used to analyze the relative risks of re-hospitalizations, between groups over follow-ups. Content analysis will be conducted for qualitative interview data.

Expected results: The PASIM is the first peer-supported self-help for illness management intervention for early-stage psychosis, particularly in Chinese population. It can be a useful and potential cost-saving intervention in community mental healthcare service, providing accessible, self-learned illness self-management training facilitated by peer-support workers (persons recovered from psychosis) in views of limited healthcare resources and mental health professionals in locally and internationally.

ELIGIBILITY:
Inclusion Criteria:

* Primarily diagnosed with psychosis (or ROP with <5 years of illness as defined in recent literature), including brief, first-episode and other psychotic disorders according to the criteria of the DSM-5 [American Psychiatric Association 2013];
* H.K. Chinese residents, aged 18-64 years;
* Global Assessment of Functioning scores ≥51, indicating mild to moderate symptoms and difficulties in psychosocial/occupational functioning [American Psychiatric Association 2013], being mentally stable to comprehend APSI or psychoeducation and outcome measures;
* Able to read and understand Cantonese/ Mandarin.

Exclusion Criteria:

* Have received or are receiving other psychotherapies;
* Comorbidity with other mental (learning disability, cognitive, or personality disorder) or significant medical disease(s);
* And/or communication, visual or hearing difficulty.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 186 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Patient functioning | Baseline
  The 43-item Specific Level of Functioning Scale is used to measure patient functioning across four domains: self-maintenance, social functioning, activities, and community-living skills. Each item is evaluated using a 5-point Likert scale (1=highly dependent/typical/always to 5=fully self-sufficient/never; total score range= 43-215). A higher total score indicates a higher level of functioning.
Patient functioning | Change from baseline to 1-week post-intervention
  The 43-item Specific Level of Functioning Scale is used to measure patient functioning across four domains: self-maintenance, social functioning, activities, and community-living skills. Each item is evaluated using a 5-point Likert scale (1=highly dependent/typical/always to 5=fully self-sufficient/never; total score range= 43-215). A higher total score indicates a higher level of functioning.
Patient functioning | Change from baseline to 9-month follow-up after the intervention
  The 43-item Specific Level of Functioning Scale is used to measure patient functioning across four domains: self-maintenance, social functioning, activities, and community-living skills. Each item is evaluated using a 5-point Likert scale (1=highly dependent/typical/always to 5=fully self-sufficient/never; total score range= 43-215). A higher total score indicates a higher level of functioning.
Patient functioning | Change from baseline to 18-month follow-up after the intervention
  The 43-item Specific Level of Functioning Scale is used to measure patient functioning across four domains: self-maintenance, social functioning, activities, and community-living skills. Each item is evaluated using a 5-point Likert scale (1=highly dependent/typical/always to 5=fully self-sufficient/never; total score range= 43-215). A higher total score indicates a higher level of functioning.

SECONDARY OUTCOMES:
Problem-solving ability | Baseline
  Problem-solving ability will be measured a 25-item Chinese version of Revised (Short) Social Problem-Solving Inventory. It comprises 2 domains: problem-solving style (rational, impulsive/careless and avoidance) and orientation (positive/negative). Items are rated on a 5-point Likert scale (0=not at all true to 4=extremely true; total score range= 0-100). A higher total score indicates better problem solving ability.
Problem-solving ability | Change from baseline to 1-week post-intervention
  Problem-solving ability will be measured a 25-item Chinese version of Revised (Short) Social Problem-Solving Inventory. It comprises 2 domains: problem-solving style (rational, impulsive/careless and avoidance) and orientation (positive/negative). Items are rated on a 5-point Likert scale (0=not at all true to 4=extremely true; total score range= 0-100). A higher total score indicates better problem solving ability.
Problem-solving ability | Change from baseline to the 9-month follow-up after the intervention
  Problem-solving ability will be measured a 25-item Chinese version of Revised (Short) Social Problem-Solving Inventory. It comprises 2 domains: problem-solving style (rational, impulsive/careless and avoidance) and orientation (positive/negative). Items are rated on a 5-point Likert scale (0=not at all true to 4=extremely true; total score range= 0-100). A higher total score indicates better problem solving ability.
Problem-solving ability | Change from baseline to 18-month follow-up after the intervention
  Problem-solving ability will be measured a 25-item Chinese version of Revised (Short) Social Problem-Solving Inventory. It comprises 2 domains: problem-solving style (rational, impulsive/careless and avoidance) and orientation (positive/negative). Items are rated on a 5-point Likert scale (0=not at all true to 4=extremely true; total score range= 0-100). A higher total score indicates better problem solving ability.
Psychotic symptoms | Baseline
  Psychotic symptoms will be assessed by a trained researcher using the 30-item Positive and Negative Syndrome Scale. It contains three subscales: positive symptoms, negative symptoms, and general psychopathology. Items will be rated on an 8-point scale (1= absent to 7= extreme; total score range= 30-210). A higher total score indicates more severe psychotic symptoms.
Psychotic symptoms | Change from baseline to 1-week post-intervention
  Psychotic symptoms will be assessed by a trained researcher using the 30-item Positive and Negative Syndrome Scale. It contains three subscales: positive symptoms, negative symptoms, and general psychopathology. Items will be rated on an 8-point scale (1= absent to 7= extreme; total score range= 30-210). A higher total score indicates more severe psychotic symptoms.
Psychotic symptoms | Change from baseline to 9-month follow-up after the intervention
  Psychotic symptoms will be assessed by a trained researcher using the 30-item Positive and Negative Syndrome Scale. It contains three subscales: positive symptoms, negative symptoms, and general psychopathology. Items will be rated on an 8-point scale (1= absent to 7= extreme; total score range= 30-210). A higher total score indicates more severe psychotic symptoms.
Psychotic symptoms | Change from baseline to 18-month follow-up after the intervention
  Psychotic symptoms will be assessed by a trained researcher using the 30-item Positive and Negative Syndrome Scale. It contains three subscales: positive symptoms, negative symptoms, and general psychopathology. Items will be rated on an 8-point scale (1= absent to 7= extreme; total score range= 30-210). A higher total score indicates more severe psychotic symptoms.
Insight into illness/treatment | Baseline
  Insight into illness/treatment will be assessed with the 11-item Insight and Treatment Attitude Questionnaire. Items are rated on a 3-point Likert scale (0=not necessary to receive treatment to 2=treatment should be required/continued regularly; total score range= 0-22). A higher total score indicates better insight into the illness/treatment.
Insight into illness/treatment | Change from baseline to 1-week post-intervention
  Insight into illness/treatment will be assessed with the 11-item Insight and Treatment Attitude Questionnaire. Items are rated on a 3-point Likert scale (0=not necessary to receive treatment to 2=treatment should be required/continued regularly; total score range= 0-22). A higher total score indicates better insight into the illness/treatment.
Insight into illness/treatment | Change from baseline to 9-month follow-up after the intervention
  Insight into illness/treatment will be assessed with the 11-item Insight and Treatment Attitude Questionnaire. Items are rated on a 3-point Likert scale (0=not necessary to receive treatment to 2=treatment should be required/continued regularly; total score range= 0-22). A higher total score indicates better insight into the illness/treatment.
Insight into illness/treatment | Change from baseline to 18-month follow-up after the intervention
  Insight into illness/treatment will be assessed with the 11-item Insight and Treatment Attitude Questionnaire. Items are rated on a 3-point Likert scale (0=not necessary to receive treatment to 2=treatment should be required/continued regularly; total score range= 0-22). A higher total score indicates better insight into the illness/treatment.
Rehospitalization rate | Baseline
  Rehospitalization rate will be calculated using the frequency and duration of and time to rehospitalizations over the past 5-6 months.
Rehospitalization rate | At 1-week post-intervention
  Rehospitalization rate will be calculated using the frequency and duration of and time to rehospitalizations over the past 5-6 months.
Rehospitalization rate | At 9-month follow-up after the intervention
  Rehospitalization rate will be calculated using the frequency and duration of and time to rehospitalizations over the past 5-6 months.
Rehospitalization rate | At 18-month follow-up after the intervention
  Rehospitalization rate will be calculated using the frequency and duration of and time to rehospitalizations over the past 5-6 months.
Service satisfaction | Baseline
  Service satisfaction will be assessed with the 8-item Client Satisfaction Questionnaire. Items are rated on a 4-point Likert scale (1= very dissatisfied to 4= very satisfied; total score range= 8-32). A higher total score indicates a better satisfaction with the services received/receiving.
Service satisfaction | Change from baseline to 1-week post-intervention
  Service satisfaction will be assessed with the 8-item Client Satisfaction Questionnaire. Items are rated on a 4-point Likert scale (1= very dissatisfied to 4= very satisfied; total score range= 8-32). A higher total score indicates a better satisfaction with the services received/receiving.
Service satisfaction | Change from baseline to 9- month follow-up after the intervention
  Service satisfaction will be assessed with the 8-item Client Satisfaction Questionnaire. Items are rated on a 4-point Likert scale (1= very dissatisfied to 4= very satisfied; total score range= 8-32). A higher total score indicates a better satisfaction with the services received/receiving.
Service satisfaction | Change from baseline to the 18-month follow-up after the intervention
  Service satisfaction will be assessed with the 8-item Client Satisfaction Questionnaire. Items are rated on a 4-point Likert scale (1= very dissatisfied to 4= very satisfied; total score range= 8-32). A higher total score indicates a better satisfaction with the services received/receiving.

CONTACTS AND LOCATIONS:
Overall Officials: Wai Tong Chien, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (2):
- China (2):
  - Integrated Community Centers for Mental Wellness, Hong Kong, Hong Kong
  - Psychiatric outpatient clinics in one hospital cluster of Hospital Authority, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The name and email of the researchers can be shared openly for communication and collaboration.

REFERENCES:
- [Background] Chien WT, Chong YY, Bressington D, McMaster CW. A randomized controlled trial of an acceptance-based, insight-inducing medication adherence therapy (AIM-AT) for adults with early-stage psychosis. Psychiatry Res. 2024 Sep;339:116046. doi: 10.1016/j.psychres.2024.116046. Epub 2024 Jun 17. PMID 38908265
- [Background] Chien WT, Bressington D, Lubman DI, Karatzias T. A Randomised Controlled Trial of a Caregiver-Facilitated Problem-Solving Based Self-Learning Program for Family Carers of People with Early Psychosis. Int J Environ Res Public Health. 2020 Dec 14;17(24):9343. doi: 10.3390/ijerph17249343. PMID 33327452
- [Background] Chien WT, Bressington D. A randomized controlled clinical trial of a nurse-led structured psychosocial intervention program for people with first-onset mental illness in psychiatric outpatient clinics. Psychiatry Res. 2015 Sep 30;229(1-2):277-86. doi: 10.1016/j.psychres.2015.07.012. Epub 2015 Jul 10. PMID 26193827
- [Background] Chien WT, Cheng HY, McMaster TW, Yip ALK, Wong JCL. Effectiveness of a mindfulness-based psychoeducation group programme for early-stage schizophrenia: An 18-month randomised controlled trial. Schizophr Res. 2019 Oct;212:140-149. doi: 10.1016/j.schres.2019.07.053. Epub 2019 Aug 12. PMID 31416744